CLINICAL TRIAL: NCT04182386
Title: Scandinavian Cohort Study for Optimal Use of Portal Vein Embolization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ernesto Sparrelid, Acting Head of HPB Surgery, MD PhD, Karolinska University Hospital
Other Study IDs: Scandinavian PVE study
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Neoplasm
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rPVE: Right portal vein embolization. All patients subjected to selective right portal vein embolization prior to planned hepatobiliary surgery.
  Interventions: Procedure: Portal vein embolization
- rPVE+S4: Right portal vein embolization including segment 4 portal vein branches. All patients subjected to selective right portal vein embolization including segment 4 portal vein branches prior to planned hepatobiliary surgery.
  Interventions: Procedure: Portal vein embolization

INTERVENTIONS:
Procedure: Portal vein embolization — Selective preoperative portal vein embolization

SUMMARY:
Several aspects on the use of portal vein embolization (PVE) are poorly studied and todays recommendations are based on low-grade evidence. In this Scandinavian multicenter cohort study we will study some of the controversial aspects on the use of PVE to try to provide clearer answers on its optimal use. Six tertiary university hospital hepatobiliary units in Sweden, Norway and Denmark participate and contribute with all PVE procedures performed at their units during the study period. We will then study several aspects PVE technique in relation to induced hypertrophy and surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Right-sided PVE

Exclusion Criteria:

* Left-sided PVE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scandinavian patients subjected to PVE at 6 hepatobiliary centers during the study period.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Future liver remnant hypertrophy | Based on radiology around 4 weeks before and after intervention
  Increase in future liver remnant, (%)

SECONDARY OUTCOMES:
Effect of segment 4 embolization on hypertrophy | Based on radiology around 4 weeks before and after intervention
  Increase in future liver remnant (%) dependeing on if segment 4 is embolized or not.
Effect of hyperbilirubinemia on hypertrophy | Based on radiology around 4 weeks before and after intervention
  Increase in future liver remnant (%) dependeing on the levels of bilirubin before portal vein embolization.
Effect of sarcopenia on hypertrophy | Based on radiology around 4 weeks before and after intervention
  Increase in future liver remnant (%) dependeing on the level of sarcopenia before portal vein embolization.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Sparrelid, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers on demand.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available to other researchers on demand.
Access Criteria: Data will be made available to other researchers on demand.